CLINICAL TRIAL: NCT05854823
Title: De-escalation of Postoperative Radiotherapy in Locally Advanced Head and Neck Squamous Cell Carcinoma With Pathological Complete Response/Major Pathological Response: A Single-arm, Prospective Phase II Clinical Study
Brief Title: The Efficacy and Safety of De-escalated Postoperative Radiotherapy in Locally Advanced HNSCC With pCR/MPR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fifth Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Yingpeng Peng, Director, Fifth Affiliated Hospital, Sun Yat-Sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZDWY.TJBZLK.002
Record Dates: First submitted 2023-05-03; First posted 2023-05-11 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: pathological complete response; major pathological response
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- de-escalation radiotherapy (Experimental): Postoperative radiotherapy alone
  Interventions: Radiation: dose-reduced radiotherapy

INTERVENTIONS:
Radiation: dose-reduced radiotherapy — Patients receive 50Gy/25F, 2Gy/F QD, five days a week for 5 weeks

SUMMARY:
This is an open-label, single-arm, phase II clinical trial to explore the efficacy and safety of de-escalation of postoperative radiotherapy in locally advanced head and neck squamous cell carcinoma with pathological complete response/major pathological response to neoadjuvant therapy. The eligible patients are scheduled to administered postoperative radiotherapy, PTV 50Gy/25F, instead of the standard dose of 60Gy. The overall primary study hypothesis is that reducing the dose of postoperative radiotherapy in the specific population does not affect DFS but significantly reduces treatment related adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Untreated, histologically confirmed head and neck squamous cell carcinoma (oral cavity, oropharynx, hypopharynx or larynx), staging T3-4N0M0 or T1-4N1-3M0, III-IVB, according to the eighth edition of the AJCC staging system; within 6 weeks after receiving neoadjuvant therapy and radical surgery.
2. Pathological evaluation of surgical specimens was pCR (pathologic complete response, no viable tumor cells) or MPR (Major pathologic response, residual viable tumor cells≤10%).
3. Negative surgical margin.
4. No extranodal extension.
5. Aged ≥ 18 years and ≤ 70 years.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
7. Life expectancy of more than 6 months.
8. Adequate organ function, based on meeting all of the following criteria (no blood components and cytologic growth factors were received within 14 days prior to the test):

   1. Hemoglobin ≥ 75 g/L; absolute neutrophil count ≥ 1.5 × 10^9/L; and platelet count ≥ 100 × 10^9/L;
   2. Serum albumin ≥ 25 g/L;
   3. Total bilirubin ≤ 1.5 × upper limit of normal (ULN); ALT and AST ≤ 2.5 × ULN;
   4. Serum creatinine ≤ 1.5 × ULN;
   5. Activated partial clotting enzyme time and international standardized ratio (INR) ≤ 1.5 × ULN (Patients on stable doses of anticoagulant therapy such as low molecular weight heparin or warfarin with INR within the expected treatment range of anticoagulants can be screened ).
9. Women of childbearing age should agree to the use of contraception (e.g., intrauterine devices, birth control pills, or condoms) during treatment and for 3 months thereafter.
10. The regimen of neoadjuvant therapy can be determined by the clinician.
11. Subjects voluntarily join the study and sign an informed consent form, with good compliance.

Exclusion Criteria:

1. Pregnant or lactating women.
2. A history of other malignant tumors within the previous 5 years or at the time of enrollment, except for cured skin basal cell carcinoma and cervical in situ cancer, as well as thyroid papilloma.
3. Neoadjuvant therapy or radical surgery was not completed.
4. Recurrence or distant metastasis occurred before postoperative radiotherapy.
5. There are contraindications for radiotherapy, chemotherapy, immunotherapy and targeted therapy.
6. Uncontrolled cardiac clinical symptoms or diseases.
7. Serious infections.
8. A history of immunodeficiency, including HIV-positive status or other acquired congenital immunodeficiency diseases, or a history of organ transplantation and bone marrow transplantation.
9. Patients with active tuberculosis infection found by history or CT examination, or patients with active tuberculosis infection history within 1 year prior to enrollment, or patients with active tuberculosis infection history before 1 year without formal treatment.
10. Active hepatitis B (HBV DNA ≥ 2,000 IU/mL or 10,000 copies/mL) or hepatitis C (positive HCV antibody test and HCV RNA above the lower limit of detection).
11. Known history of psychotropic drug abuse, alcoholism and drug use.
12. Not suitable for inclusion, as judged by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2023-04-10 (Actual); Primary Completion 2027-04-09 (Estimated); Study Completion 2027-04-09 (Estimated)

PRIMARY OUTCOMES:
Disease Free Survival (DFS) | from the first day of treatment to the follow up of 2 years
  2-year disease free survival rate

SECONDARY OUTCOMES:
Overall Survival (OS) | from the first day of treatment to the follow up of 2 years
  2-year overall survival rate
Local Relapse Free Survival (LRFS) | from the first day of treatment to the follow up of 2 years
  2-year local relapse free survival rate
Distant Metastasis Free Survival (DMFS) | from the first day of treatment to the follow up of 2 years
  2-year distant metastasis free survival rate
EORTC QLQ-C30 | from 1 week before treatment to the follow up of 2 years
  Quality of life evaluation
EORTC HN35 | from 1 week before treatment to the follow up of 2 years
  Quality of life evaluation
RTOG/EORTC late radiation morbidity scoring scheme | from 1 week before treatment to the follow up of 2 years
  Toxicity criteria of RTOG/EORTC

CONTACTS AND LOCATIONS:
Locations (1):
- Fifth Affiliated Hospital of Sun Yat-sen University, Zhuhai, Guangdong, China